CLINICAL TRIAL: NCT04879108
Title: The Role of Transcutaneous Electrical Nerve Stimulation Combined With Physiotherapy and Rehabilitation Program on Pulmonary Function and Functional Exercise Capacity in Patients Undergoing Thoracic Surgery? A Randomized Controlled Trial
Brief Title: The Effectiveness of Transcutaneous Electrical Nerve Stimulation After Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 5563
Record Dates: First submitted 2021-05-02; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Thoracic; Surgery; Pain; Pulmonary Function; Functional Capacity
Keywords: transcutaneous electrical nerve stimulation; physiotherapy and rehabilitation; thoracic surgery; pain; pulmonary function; functional capacity
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Crossover Assignment Randomized controlled
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor (pain, pulmonary function tests, 6 minute walking test, peak cough flow)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy rehabilitation and Transcutaneous Electrical Nerve Stimulation (TENS) group (Experimental): Physiotherapy rehabilitation and Transcutaneous Electrical Nerve Stimulation (TENS) group received TENS therapy in addition to physiotherapy rehabilitation approaches after thoracic surgery.
  Physiotherapy and rehabilitation program was started after surgery and it was performed for 30 min, twice a day, 5 day a week. The program was included respiratory and posture exercises, coughing, enhancing mobility.
  TENS therapy was performed with the a 2-channel portable TENS device and using disposable electrodes. TENS applied on both sides of the incision line. After surgery, TENS was performed before the Physiotherapy rehabilitation for 30 min, twice a day, 5 day a week.
  Patients were evaluated before the surgery and the end of postoperative 5th day.
  Interventions: Other: Physiotherapy rehabilitation and Transcutaneous Electrical Nerve Stimulation
- Physiotherapy rehabilitation Group (Active Comparator): This group was enrolled only physiotherapy and rehabilitation program after thoracic surgery.
  Physiotherapy and rehabilitation program was started after surgery and it was performed for 30 min, twice a day, 5 day a week. The program was included respiratory and posture exercises, coughing, enhancing mobility.
  Patients were evaluated before the surgery and the end of postoperative 5th day.
  Interventions: Other: Physiotherapy Rehabilitation

INTERVENTIONS:
Other: Physiotherapy rehabilitation and Transcutaneous Electrical Nerve Stimulation — Physiotherapy rehabilitation and Transcutaneous Electrical Nerve Stimulation (TENS) group received TENS therapy in addition to physiotherapy rehabilitation after thoracic surgery.
  Physiotherapy and rehabilitation program was started after surgery and it was performed for 30 min, twice a day, 5 day a week. The program was included respiratory and posture exercises, coughing, enhancing mobility.
  Transcutaneous Electrical Nerve Stimulation was performed with the a 2-channel portable TENS device and using disposable electrodes. TENS applied on both sides of the incision line. After surgery, TENS was performed before the Physiotherapy and Rehabilitation for 30 min, twice a day, 5 day a week.
  Patients were evaluated before the surgery and the end of postoperative 5th day.
  Arms: Physiotherapy rehabilitation and Transcutaneous Electrical Nerve Stimulation (TENS) group
Other: Physiotherapy Rehabilitation — Physiotherapy and Rehabilitation was performed for 5 days after surgery, twice a day, for 30 min, 5 day a week after thoracic surgery. The program was included respiratory and posture exercises, coughing, enhancing mobility.
  Patients were evaluated before the surgery and the end of postoperative 5th day.
  Arms: Physiotherapy rehabilitation Group

SUMMARY:
The purpose of this randomised and controlled study is to investigate the effects of transcutaneous electrical nerve stimulation combined with physiotherapy and rehabilitation program on pulmonary function and functional exercise capacity.

DETAILED DESCRIPTION:
Post-thoracotomy pain is one of the most severe types of post-surgical pain. When pain after thoracotomy is not treated effectively, it causes decrease in pulmonary compliance, inability to cough and deep breathing. Increased secretion leads to atelectasis and pneumonia. After surgery, early mobilization, providing airway cleaning (humidification, aspiration, forced expiration, assisted coughing), oxygen therapy, controlled breathing exercises, the use of incentive spirometry and such selected exercises, including posture and general exercises physiotherapy and rehabilitation approaches can prevent complications. A carefully planned pre and postoperative chest physiotherapy and rehabilitation program minimizes postoperative complications; it will restore normal function in these patients. Post-surgical physiotherapy applications should be combined with pain therapy for effective participation of the patient.

Local anesthetics, opioids and different special analgesia techniques including intercostal, paravertebral, interpleural and epidural blocks are used to relieve pain after thoracotomy. However, these techniques have serious side effects such as nausea, vomiting, respiratory depression, and sleepiness. It has been reported that the use of Transcutaneous Electrical Nerve Stimulation (TENS), in addition to traditional analgesia methods, may reduce the use of analgesics, side effects, and postoperative recovery period, and is useful for pain control. After cardiac surgery, TENS has been found useful in the treatment of postoperative incision pain. It has been reported that TENS therapy after thoracotomy as effective as patient-controlled analgesia.

Therefore, this study planned to investigate the effects of transcutaneous electrical nerve stimulation combined with physiotherapy and rehabilitation program on pulmonary function and functional exercise capacity in patients undergoing thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lobectomy for lung cancer

Exclusion Criteria:

* Patients undergoing pneumonectomy.
* Patients undergoing smaller resection than lobectomy.
* Presence of serious arrhythmia, pacemaker, severe cardiac failure,
* Patients with cooperation disorder
* Presence of neurological or orthopedic problems affecting the extremities.
* Patients with severe psychiatric disorders

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2011-04-30 (Actual); Study Completion 2011-09-05 (Actual)

PRIMARY OUTCOMES:
Functional Exercise Capacity | Change from Baseline Functional Exercise Capacity at postoperative 5th days.
  Functional exercise capacity was measured with the 6 Minute Walk Test according to the American Thoracic Society guidelines. The 6 minutes walking distance was recorded in meters.
Forced expiratory volume in one second Spirometric measurement | Change from Baseline Functional Exercise Capacity at postoperative 5th days.
  Forced expiratory volume in one second spirometric measurement was measured. Test was carried out according to American Thoracic Society / European Respiratory Society criteria.
Forced Vital Capacity Spirometric measurement | Change from Baseline Functional Exercise Capacity at postoperative 5th days.
  Forced Vital Capacity spirometric measurement was measured. Test was carried out according to American Thoracic Society / European Respiratory Society criteria.
Pain severity | Baseline and postoperative 5th days.
  Visual Analogue Scale that is an easy, reproducible, minimal tool-requiring, and understandable measurement tool for the assessment of pain intensity was used. This scale consists of a horizontal, straight line. There is a value of 0 at the beginning of the line and 10 at the end.
Peak cough flow | Change from Baseline Functional Exercise Capacity at postoperative 5th days.
  It was evaluated with the peak flow meter device while the patient was sitting upright in a chair with a back. The test method is explained and a trial test is carried out. The nosepiece was attached to the nose and the mouthpiece of the device was wrapped tightly with the lips.
  It was asked to take a deep breath and suddenly and quickly blow into the device fron the patient. The best out of three acceptable tests was recorded.

SECONDARY OUTCOMES:
Evaluation of dyspnea | Baseline and postoperative 5th days.
  It was evaluated with a 0-10 point borg scale. Dyspnea was measured at rest and after exertion. An increase in score is interpreted as an increase in dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Yildiz Ozer, PT, PhD, Principal Investigator — Marmara University; Nilgun Gurses, Prof, Study Director — Bezmialem Vakif University; Alper Toker, Prof, Study Chair — Istanbul University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Erdogan M, Erdogan A, Erbil N, Karakaya HK, Demircan A. Prospective, Randomized, Placebo-controlled Study of the Effect of TENS on postthoracotomy pain and pulmonary function. World J Surg. 2005 Dec;29(12):1563-70. doi: 10.1007/s00268-005-7934-6. PMID 16331341
- [Result] Cesario A, Ferri L, Galetta D, Pasqua F, Bonassi S, Clini E, Biscione G, Cardaci V, di Toro S, Zarzana A, Margaritora S, Piraino A, Russo P, Sterzi S, Granone P. Post-operative respiratory rehabilitation after lung resection for non-small cell lung cancer. Lung Cancer. 2007 Aug;57(2):175-80. doi: 10.1016/j.lungcan.2007.02.017. Epub 2007 Apr 17. PMID 17442449
- [Result] Kaneda H, Saito Y, Okamoto M, Maniwa T, Minami K, Imamura H. Early postoperative mobilization with walking at 4 hours after lobectomy in lung cancer patients. Gen Thorac Cardiovasc Surg. 2007 Dec;55(12):493-8. doi: 10.1007/s11748-007-0169-8. Epub 2007 Dec 11. PMID 18066640
- [Result] Benedetti F, Amanzio M, Casadio C, Cavallo A, Cianci R, Giobbe R, Mancuso M, Ruffini E, Maggi G. Control of postoperative pain by transcutaneous electrical nerve stimulation after thoracic operations. Ann Thorac Surg. 1997 Mar;63(3):773-6. doi: 10.1016/s0003-4975(96)01249-0. PMID 9066400
- [Result] Sancho J, Servera E, Diaz J, Marin J. Comparison of peak cough flows measured by pneumotachograph and a portable peak flow meter. Am J Phys Med Rehabil. 2004 Aug;83(8):608-12. doi: 10.1097/01.phm.0000133431.70907.a2. PMID 15277962
- [Result] Meek PM. Measurement of dyspnea in chronic obstructive pulmonary disease: what is the tool telling you? Chron Respir Dis. 2004;1(1):29-37. doi: 10.1191/1479972304cd008ra. PMID 16281665
- [Result] Freynet A, Falcoz PE. Is transcutaneous electrical nerve stimulation effective in relieving postoperative pain after thoracotomy? Interact Cardiovasc Thorac Surg. 2010 Feb;10(2):283-8. doi: 10.1510/icvts.2009.219576. Epub 2009 Nov 12. PMID 19910359